CLINICAL TRIAL: NCT02266654
Title: Early Goal Directed Therapy in Sepsis by EMS
Brief Title: Early Goal Directed Therapy in Sepsis by Emergency Medical Services
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll participants
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Pro EMS (Unknown); Mount Auburn Hospital (Other)
Responsible Party: Principal Investigator, Michael Filbin, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 019-2014
Record Dates: First submitted 2014-06-09; First posted 2014-10-17 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Sepsis
Keywords: Emergency Medical Services; Lactic Acid; Sepsis
MeSH Terms: conditions — Sepsis | interventions — Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prehospital-directed therapy arm (Experimental): Patients who are hypotensive or whose lactate is ≥ 2.5, prehospital providers will provide a notification to the receiving hospital (Hospital Notification), establish an IV, and provide 1 liter normal saline (NS) bolus of IV fluids. An additional 1 liter normal saline bolus will be given for systolic blood pressure less than 100. Patients who have a history of end-stage renal disease or congestive heart failure would receive only 20 milliliters/kilogram of fluid. If the patient remains hypotensive, Emergency Medical Services will continue providing fluids as is standard of care.
  Interventions: Other: IV fluids; Other: Hospital Notification
- Control Arm (Experimental): Prehospital providers will obtain a point of care lactate, establish an IV, and provide IV fluids as judged necessary.
  Interventions: Other: IV fluids

INTERVENTIONS:
Other: IV fluids — Normal Saline 0.9%
Other: Hospital Notification — Prehospital providers will notify the receiving hospital over the radio or telephone that they are transporting a patient who meets Sepsis Criteria
  Arms: Prehospital-directed therapy arm

SUMMARY:
The goal is to evaluate the best way for paramedics and hospitals to work together to treat septic patients as quickly as possible.

The investigators think that the best thing to do for septic patients is to identify and treat them as early as possible. This research will test this. The investigators think that if paramedics identify septic patients and begin treatment with fluids in the ambulance, then the patient will do better in the long run. The paramedic will also tell the hospital that a septic patient will be there soon. The caregivers can prepare and be ready to provide care as soon as the patient arrives. With this research, the investigators would like to see if these steps help patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years of age
* Suspected to having an infection
* Meets 2 of 3 systemic inflammatory response criteria: heart rate > 90 beats per minute, respiratory rate >20 breaths per minute, temperature >38°C or <36°C

Exclusion Criteria:

* Transfer from another hospital
* Patients, coming from a rehabilitation/nursing facility where antibiotics were given prior to transfer
* Pregnant patients
* Prisoners.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Time to antibiotics | During the Emergency Department stay (expected to be 5 hours)

SECONDARY OUTCOMES:
Mortality | Participants will be followed for the duration of hospital stay, an expected average of 1 week
Need for pressors in the Emergency Department | During the Emergency Department stay (expected to be 5 hours)
Admitted to the Intensive Care Unit from the Emergency Department | During the Emergency Department stay (expected to be 5 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Filbin, MD, Principal Investigator — Massachusetts General Hospital; William Porcaro, MD, MPH, Principal Investigator — Mount Auburn Hospital
Locations (1):
- Mount Auburn Hospital, Cambridge, Massachusetts, United States